CLINICAL TRIAL: NCT00411372
Title: A Randomized, Double-blind, Parallel-group Study of Fluticasone Propionate/Salmeterol Combination (FSC 250/50mcg) Twice Daily and Salmeterol (SAL 50mcg) Twice Daily to Validate a New Shortness of Breath Questionnaire in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Shortness Of Breath Questionnaire Validation Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No subjects enrolled. Study was canceled before active
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCO105782
Record Dates: First submitted 2006-12-13; First posted 2006-12-14 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Questionnaire; COPD; Shortness of Breath
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Fluticasone; Salmeterol Xinafoate

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol 250/50mcg combination, salmeterol 50mcg
  Other Names: fluticasone propionate/salmeterol 250/50mcg combination; salmeterol 50mcg

SUMMARY:
This study will last for approximately 8 weeks and will involve 4 visits. The study is being carried out to validate a shortness of breath questionnaire

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of COPD

Exclusion Criteria:

* Women who are pregnant or lactating.
* Subjects with a primary diagnosis of asthma. (Subjects with a prior history of asthma are eligible if COPD is currently their primary diagnosis)
* Has a respiratory disorder other than COPD (e.g., bronchiectasis, sarcoidosis, active tuberculosis, lung fibrosis), including subjects with a diagnosis of alpha-1-antitrypsin deficiency.
* Subjects with lung volume reduction surgery or lung transplant within the previous 12 months.
* Chest X-ray (posterior-anterior) or CT scan reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD. A chest X-ray must be taken if the subject has not had one within 12 months of the Screening Visit.
* Subjects with clinically significant cardiovascular (including clinically significant ECG abnormalities, CHF), neurological, psychiatric, renal, immunological, endocrine(including uncontrolled diabetes or thyroid disease) or hematological abnormalities that is uncontrolled.
* Subjects with carcinoma that has not been in complete remission for at least 5 years. Carcinoma in situ of the cervix, squamous cell carcinoma of the skin and basal cell carcinoma would not be considered exclusion criteria if the subject was considered cured in less than 5 years since diagnosis.
* Any adverse reaction including immediate or delayed hypersensitivity to any betaagonist, sympathomimetic drug, or intranasal, inhaled, or oral corticosteroid including any components of the formulations (e.g. lactose or milk protein).
* Initiation of systemic beta-blocker medications at any time during the study. Systemic beta-blockers and beta-blocker eye drops are allowed for those subjects who have been on a stable regimen for at least 30 days prior to screening and judged capable to continue this regimen until discharged from the study.
* Subject continues on any prohibited medications, as listed in Section 5.6.2.
* Subject is receiving treatment with long-term oxygen therapy (LTOT), defined as inSection 5.6.2.
* Use of immunosuppressive medications at any time during the study. Immunotherapy for the treatment of allergies is allowed during the study provided that the subject has received a constant dose for 30 days prior to the Screening Visit and the dose is maintained during the study.
* Subjects who are medically unable to withhold their albuterol or ipratropium for the 6 hour period required prior to administration of questionnaires and spirometry at each study visit.
* An infection of the upper or lower respiratory tract requiring treatment with antibiotics 14 days prior to the Screening Visit.
* Subjects who require nocturnal positive pressure.
* Enrolled in or discontinuation of a pulmonary rehabilitation program within 30 days of Visit 1. Subjects who are enrolled in a pulmonary rehabilitation program at study start should maintain participation in the program for the duration of the study.
* Use of any investigational drug within 30 days of Visit 1 or at any time during the study is not allowed.
* Subjects unable to comply with study procedures.
* Study investigators, sub-investigators, study coordinators, employees of a participating investigator or immediate family members of the aforementioned are excluded from participation in this study.
* Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation, substance abuse, (including drug and alcohol), or other conditions, which will limit the validity of informed consent to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11

PRIMARY OUTCOMES:
The objective of this study is the validation of the Shortness of Breath Questionnaire in subjects with COPD

SECONDARY OUTCOMES:
spirometry (FEV1, FVC, IC)
diary card data
Health Outcomes (Chronic Respiratory Questionnaire - SAS, Clinical Global Impression of Dyspnea Severity, Patient Global Assessment of Change Question, Clinical Global Impression of Change Question

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline